CLINICAL TRIAL: NCT05858671
Title: Determining the Lipid Lowering Effect of Fenugreek Seed Tea: a Randomized Controlled Trial
Brief Title: Determining the Lipid Lowering Effect of Fenugreek Seed Tea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Jayne Woodside, PhD, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20/NI/0057
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Hyperlipidemias
Keywords: Fenugreek; Hyperlipidaemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Tea

STUDY DESIGN:
Intervention Model Description: This will be a randomised controlled trial. 114 participants will be randomized into two groups (57/group) to receive either fenugreek seed tea or a control black tea, respectively.
Who Masked: Participant
Masking Description: The study will be single blind as the participants will not know to what treatment they have been allocated until the end of the study. However, as the Postdoctoral Research Fellow will be conducting study visits and allocating participants to their treatment group it will not be possible for them to be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fenugreek Seed Tea (Experimental): Fenugreek seeds will be delivered at a dose of 5g/day, drunk as a tea (2.5g/per tea bag), p.o. twice a day at a 12-hour interval) for 8 weeks (56 days). The tea bags will be brewed in a cup (200ml) of boiled hot water for 10 minutes before drinking. This will be self-administered by the subjects, twice a day at a 12-hour interval. The rationale for choosing the dose and intervention time course were based on the previous studies where metabolic effects have been detected. Literature reports from 12 human studies on diabetic and pre-diabetic subjects gave doses of fenugreek seed ranging from 1 to 100g/day, with the median treatment dose being 6.3g/day, to the participants; the intervention time course ranged from 1 week to 3 years, with the median treatment time being 60 days. The dose and duration in this study was designed as being similar to these studies where metabolic effects have been detected and where participant burden will not be too onerous.
  Interventions: Other: Fenugreek Seed Tea
- Black Tea (Placebo Comparator): Control group: A control black tea (2.5g/bag), self-administered by the subjects, twice in a day at a 12-hour interval. Black tea is a type of fermented tea that has been found to possess much less cardioprotective and lipid profile improving effect compared to green tea due to the different manufacture process. Consumption of black tea has been found not associated with a reduced risk of coronary heart disease in the United Kingdom. Therefore, we propose to use black tea as control tea for this study.
  Interventions: Other: Black Tea

INTERVENTIONS:
Other: Fenugreek Seed Tea — Fenugreek seeds will be delivered at a dose of 5g/day, drunk as a tea (2.5g/per tea bag), p.o. twice a day at a 12-hour interval) for 8 weeks (56 days). The tea bags will be brewed in a cup (200ml) of boiled hot water for 10 minutes before drinking. This will be self-administered by the subjects, twice a day at a 12-hour interval.
  Arms: Fenugreek Seed Tea
Other: Black Tea — A control black tea (2.5g/bag), self-administered by the subjects, twice in a day at a 12-hour interval.
  Arms: Black Tea

SUMMARY:
The goal of this randomized clinical trial is to investigate the lipid-lowering effect of fenugreek seed consumed as a tea in patients with hyperlipidaemia, but without diabetes over an 8-week intervention period. Alteration of plasma microRNAs (e.g. microRNA-122 and microRNA-34a) will further be analysed for establishing as non-invasive therapeutic biomarkers of hyperlipidaemia. Participants will be asked to attend three study at baseline, 4 and 8 weeks in the Centre for Public Health. Each visit will involve the collection of demographic information, anthropometric measurements, blood pressure and fasting blood samples. Participants allocated to intervention or control will be asked to self-administer tea twice a day at a 12 hour interval over the 8-week study period. Researchers will compare the results of the consumption of fenugreek seed tea to the control black tea to see if fenugreek has any effect on lipid levels.

DETAILED DESCRIPTION:
Poor regulation of lipid metabolism and hyperlipidemia are central to the development of cardiovascular disease (CVD). Hyperlipidemia is characterized as the overproduction of very low density cholesterol and low density lipoprotein (LDL) (i.e. bad cholesterol) and decreased high density lipoprotein (HDL) (i.e. good cholesterol). Amongst individuals with mild to moderate hyperlipidemia, lifestyle changes is the first treatment option, such as a healthy diet. Therefore, seeking to develop food-based approaches for hyperlipidemia therapy is a timely endeavour. Fenugreek has been suggested as an attractive option, as it is a spice throughout the world which possesses medicinal properties in regulating human nutrient metabolism. In a recent review of the overall effects of fenugreek on hyperlipidemia in humans with diabetes and prediabetes, this analysis suggested that fenugreek has total cholesterol-lowering efficacy. The effects of fenugreek on triglyceride and LDL-cholesterol showed a trend towards reduction and an incremental trend for HDL-cholesterol but needed further confirmation. The effect of fenugreek in human subjects with hyperlipidemia without diabetes has not been investigated. This research aims to investigate the lipid-lowering effect of fenugreek seed consumed as a tea in patients with hyperlipidaemia, but without diabetes over an 8-week intervention period. Changes in plasma microRNAs will be analysed to establish non-invasive therapeutic biomarkers of hyperlipidemia.

Participants without pre-existing CVD or diabetes aged 18-70 years old will be included if they have hyperlipidemia (plasma triglyceride level between 1.7 - 4.5mmol/l) not on any lipid-lowering treatment or on a stable lipid-lowering treatment (last six months) but still have confirmation of high triglycerides within the range required for study.

114 participants will be randomized into two groups (57/group) to receive either fenugreek seeds or control tea, respectively. Treatment allocations will be placed into sealed envelopes and this will be opened at the baseline study visit with the participant.

Fenugreek seeds will be delivered at a dose of 5g/day, drunk as a tea (2.5g/per tea bag), p.o. twice a day at a 12-hour interval) for 8 weeks (56 days). The tea bags will be brewed in a cup (200ml) of boiled hot water for 10 minutes before drinking. This will be self-administered by the subjects, twice a day at a 12-hour interval. The rationale for choosing the dose and intervention time course were based on the previous studies where metabolic effects have been detected. Literature reports from 12 human studies on diabetic and pre-diabetic subjects gave doses of fenugreek seed ranging from 1 to 100g/day, with the median treatment dose being 6.3g/day, to the participants; the intervention time course ranged from 1 week to 3 years, with the median treatment time being 60 days. The dose and duration in this study was therefore designed as being similar to these studies where metabolic effects have been detected, and also, where participant burden will not be too onerous, at a dose of 5g/day, twice a day at a 12-hour interval for 8 weeks (56 days). For the control group, a control black tea (2.5g/bag), self-administered by the subjects, twice in a day at a 12-hour interval. Black tea is a type of fermented tea that has been found to possess much less cardioprotective and lipid profile improving effect compared to green tea due to the different manufacture process. Consumption of black tea has been found not associated with a reduced risk of coronary heart disease in the United Kingdom.

Recruitment will be via outpatient hyperlipidemia clinics, primary care and advertisements. Study visits will take place at the Centre for Public Health at baseline, 4 and 8 weeks and will involve the collection of demographic information, anthropometric measurements, blood pressure and fasting blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients aged between 18-70 years old
* Patients with hyperlipidaemia (plasma triglyceride level between 1.7 - 4.5mmol/l) not on any lipid-lowering treatment or on a stable lipid-lowering treatment (last six months) but still have confirmation of high triglycerides within the range required for study
* Willing not to change any dietary behaviours, with the exception of participating in the intervention, over the course of the study
* Participants can be recruited onto the study if they are involved in other research studies, but this will depend on the study type and the decision will be made by the Chief Investigator and/or Principal Investigator.

Exclusion Criteria:

* Patients with type 1 or type 2 diabetes, asthma, allergic reactions, respiratory, kidney, and neurological diseases, psychiatric disorders or pre-existing CVD
* Living in a residential or nursing care home
* Taking high dose nutritional supplements above the dietary reference values
* Consumption of alcohol above current recommended levels (14 units per week), pregnancy or lactation
* Inability to provide informed consent
* Any other problem which would prevent adherence to fenugreek intervention

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Serum triglycerides | 8 weeks
  The primary outcome of this study is between group differences in mean change in serum triglycerides.

SECONDARY OUTCOMES:
Total-cholesterol | 8 weeks
  Between group differences in mean change in total-cholesterol
LDL-cholesterol | 8 weeks
  Between group differences in mean change in LDL-cholesterol
non-HDL-cholesterol | 8 weeks
  Between group differences in mean change in non-HDL-cholesterol
HDL-cholesterol | 8 weeks
  Between group differences in mean change in HDL-cholesterol
Plasma apolipoprotein B | 8 weeks
  Between group differences in mean change in plasma apolipoprotein B, whose level reflects plasma very low-density lipoprotein (VLDL) contents
MicroRNAs | 8 weeks
  Between group differences in mean changes of plasma microRNA-122 and microRNA-34a as non-invasive therapeutic biomarkers in human subjects involved in this study

CONTACTS AND LOCATIONS:
Overall Officials: Jayne Woodside, PhD, Principal Investigator — Queen's University, Belfast
Locations (2):
- United Kingdom (2):
  - Centre for Public Health, Institute of Clinical Sciences A, Belfast, Northern Ireland
  - Queen's University Belfast, Belfast

IPD SHARING:
Plan to Share IPD: Yes
The researchers are happy to share results from the study for the purposes of a meta-analysis. This will be completed on approach to the researchers.
Supporting Information: Study Protocol, ICF
Time Frame: Data should be available from June 2024 and will be available for 2 years.
Access Criteria: Use of results in a meta-analysis.